CLINICAL TRIAL: NCT00533728
Title: A Phase I Study to Determine the Safety and Effect of Soluble Beta-Glucan (SBG) in Combination With Rituximab and COP/CHOP in Patients With Non'Hodgkin's Lymphoma
Brief Title: Safety of Soluble Beta-Glucan (SBG) in Treatment of Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biotec Pharmacon ASA (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBG-2-02
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2009-03-04 (Estimated); Status verified 2009-03

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Soluble beta-glucan (SBG)

SUMMARY:
The purpose of this study is to assess the safety of soluble beta-glucan (SBG) in combination with antibody and chemotherapy treatment in patients with non-Hodgkin-s lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. CD20 positive B-cell non-Hodgkin's lymphoma
2. Treatment with rituximab and CHOP or COP
3. Performance status 0 or 1 according to the WHO scale (Appendix)
4. Expected lifetime of more than 12 weeks
5. Age ≥ 18 years
6. The patient must be able and willing to comply with the study procedures, and signed and dated informed consent must be obtained

Exclusion Criteria:

1. Women who are pregnant or breast-feeding. For fertile women, a negative pregnancy test must be provided during the screening test. Women of childbearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation
2. Lymphoma involvement of central nervous system
3. Reduced bone marrow function defined by leukocyte counts < 3.0 x 109/l, neutrophil counts < 1.5 x 109/l, thrombocyte counts < 100 x 109/l or hemoglobin < 10 g/dl
4. Reduced liver function defined by bilirubin > 1.5 x upper limit of normal (ULN) or ASAT/ALAT ≥ 3 x ULN
5. Reduced renal function defined by serum creatinine ≥ 2 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Lehne, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Rikshospitalet, Kreftklinikken Radiumhospitalet, Oslo, Norway